CLINICAL TRIAL: NCT04113486
Title: Expression Levels of Nicotinamide Metabolism-related Protein (NMAP) in Newly Diagnosed Renal Cancer and Non-renal Cancer Populations
Acronym: ENRC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jie Ding, Attending doctor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2019-104
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cancer; tumor biomarker
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Renal cancer group: Patients which imaging studies have found renal mass, plan to receive surgery (except for radiofrequency ablation, cryoablation, etc.), about 100.
  Interventions: Other: Blood test
- Urothiasis group: Patients which imaging studies have found renal or ureteral stones, and rule out of renal mass, about 100.
  Interventions: Other: Blood test
- Renal cysts group: Patients which imaging studies have found renal cysts (simple or complex) about 100.
  Interventions: Other: Blood test
- Liver cancer group: Patients which imaging studies have found hepatic mass, plan to receive surgery (except for radiofrequency ablation, cryoablation, etc.), about 100.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — About 4 ml of blood draw

SUMMARY:
This study aims to observe the difference between NMAP (nicotinamide metabolism associated protein) serum levels in primary diagnosed renal cancer patients and non-renal cancer patient controls, plot the ROC curve and establish appropriate cut-off values.

ELIGIBILITY:
Inclusion Criteria:

1. The tumor group patients were found to have renal or hepatic mass, plan to receive surgical treatment (except for radiofrequency ablation, cryoablation, etc., which were not available for pathological examination). The control group patients were ruled out of tumor based on radiological tests and commonly used tumor biomarkers
2. Age ≥ 18 years old and able to provide written informed consent;
3. Have not received any systemic or topical treatment for kidney/liver tumors.
4. Cardiopulmonary, liver and kidney functions are able to tolerate surgery and can comply with research requirements.

Exclusion Criteria:

1. The investigators believe that the subject may be unsuitable for inclusion due to severe concurrent diseases, infections, and etc.
2. The subjects is known or suspected of other malignancies.
3. There has been another history of malignancy in the past 5 years.
4. Major surgery (surgery requiring general anesthesia) was performed within 4 weeks prior to screening visits.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients are in-hospital patients treated in Xinhua Hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
NMAP level study | September 2019-September 2021
  To observe the difference in the expression level of nicotinamide metabolism related protein (NMAP) in the serum of newly diagnosed renal cancer and non-renal cancer patients. Draw the NMAP ROC curve and establish the appropriate Cut-off value to analyze its sensitivity and specificity.

SECONDARY OUTCOMES:
NMAP plus other tumor biomarkers study | September 2019-September 2021
  According to NMAP and combined with other tumor biomarkers data such as AFP, multiple regression analysis was used to map the ROC curve and establish the appropriate Cut-off value to determine whether it is capable of distinguishing kidney cancer and liver cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to reveal IPD due to further research plan